CLINICAL TRIAL: NCT02604173
Title: A Randomized Controlled Trial of Altitude Sickness Prevention and Efficacy of Comparative Treatments
Brief Title: Altitude Sickness Prevention and Efficacy of Comparative Treatments
Acronym: ASPECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Associate Professor Department of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 35330
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Budesonide; Acetazolamide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Budesonide (Experimental): Budesonide inhaler as experimental treatment along with placebo pill.
  Interventions: Drug: Budesonide
- Acetazolamide (Active Comparator): Acetazolimide pill as active comparator along with sham inhaler.
  Interventions: Drug: Acetazolamide
- Control (Sham Comparator): Sham inhaler as control for budesonide inhaler along with placebo pill as control for acetazolamide comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Inhaled Budesonide vs. PO Acetazolamide vs. Placebo for prevention of Acute Mountain Sickness
  Other Names: entocort, pulmicort
  Arms: Budesonide
Drug: Acetazolamide — Inhaled Budesonide vs. PO Acetazolamide vs. Placebo for prevention of Acute Mountain Sickness
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Placebo — Placebo pill and sham inhaler
  Other Names: sugar pill
  Arms: Control

SUMMARY:
This study is designed to be the first to examine the novel drug budesonide for prevention of acute mountain sickness in comparison to acetazolamide and in the context of rapid ascent to high altitude. The investigators will accomplish these objectives with a prospective, double blinded view of a large population of hikers who are ascending at their own rate in a true hiking environment.

DETAILED DESCRIPTION:
Enrollment:

A total of One hundred healthy male and female participants (group of 25 at a time) will be enrolled by study administrators at Owens Valley Lab, White Mountain Research Station. Pregnant women will be excluded. The study enrollment period will run for approximately 12 days over 4 weekends in August 2016. Advertisement of the study at sea level locals in and around Stanford University as well as email chains with other outdoor groups will attempt to gather a cohort of sea-level participants.

Study:

Eligible participants will be randomized in a double blind fashion the morning of ascent to acetazolamide 125 mg PO bid and empty inhaler, budesonide (200 mcg) inhaler bid and visually matched placebo pill, or visually matched placebo and empty inhaler. After informed consent is signed, participants will complete the baseline demographics sheet, LLQ, have pulse oximetry readings, and perform pulmonary function testing prior to taking the study medications. Participants will take the study capsules and inhaler before they leave from OVL, in order to reveal any significant acute adverse reactions before they leave for higher altitude. In the highly unlikely event of an adverse reaction, the participant will be in close proximity to study administrators who will have first aid medicines to treat allergic reactions (Benadryl, Ranitidine, Prednisone, Epinephrine), and communication to BAR where the code can be broken for medical evaluation. In the morning healthy participants without adverse reactions will drive to the Barcroft Gate 11,700', continue on foot to the Barcroft Research Station (BAR) at 12,500'. The study subjects will be allowed to hike at their own pace with minimal restrictions including no travel above 13,054' (Barcroft Summit). The participants will spend the night at BAR where they will be evaluated within 6 hours of their arrival and the morning after (LLQ, pulse oximetry, pulmonary function testing, side effects data, and compliance). After data collection the morning after arrival, the study will be completed for each participant. Participants with significant illness will be removed from the trial and appropriate safety measures taken (Twenty-four hour access to truck evacuation to lower elevations at OVL - the definitive treatment for AMS). Every effort will be made to secure the incomplete data of those who abort the study early. The highest scoring AMS data will be used for primary and secondary outcome analysis.

Procedures:

Two data collection timelines will be coordinated, one within 6 hours of subjects arrival to BAR and the second the morning after a night of sleep at BAR. Five study variables will be assessed including LLQ, pulse oximetry, pulmonary function testing, side effects data, and compliance. The LLQ is a widely used standardized self-report clinical survey used for the quantitation of AMS. A diagnosis of AMS on the LLQ requires a score of 2 or greater with the mandatory presence of headache and at least one of the following symptoms: dizziness or lightheadedness, fatigue, GI symptoms (nausea/vomiting), or difficulty sleeping. AMS symptoms are evaluated by establishing a space of time (several hours to one day normally) during which symptoms can be quantified. In this study, symptoms will be evaluated within 6 hours after arrival at the endpoint altitude, and then again the next morning to capture all those with manifestation of disease. The highest LLQ score will be used for scoring at that altitude, irrespective of an AMS diagnosis. This methodology takes into account the variable timeline for individual expression of AMS symptomatology. Oxygen saturation has a rough correlation with AMS symptoms, and will be measured with the use of a pulse oximeter, which is validated for use at high altitude (Nonin Onyx, Nonin Medical Products, Minneapolis, MN).

Pulmonary Function Testing: Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and Peak Expiratory Flow Volume (PEF). will be achieved with a portable spirometer. Values between baseline level and altitude will be computed. Spirometry will be performed according to the guidelines of the American Thoracic Society.

Side Effects Data will be recorded that the patient may be experiencing secondary to the interventions of inhaled budesonide or acetazolamide or placebo.

Compliance will be verified of whether or not the subject followed intervention guidelines through until data completion

Interventions:

Commercial pharmaceutical-grade acetazolamide will be purchased by Advantage Pharmaceuticals and will be packed in lactulose capsules by Advantage Pharmaceuticals at their processing plant in Rocklin, CA. The placebo substance will be visually identical to the acetazolamide, and both placebo and drug will be packed in visually identical capsules. Budesonide and visually identical chambers will be donated by AstraZeneca. Prior studies have established that medicated and empty inhalants are indistinguishable by study participants. The packaging of the capsules and inhalants and placebo will be randomized in a 1:1:1 strategy. The first dose to be taken at least 4 hours before ascent for up to 100 participants in three arms: placebo (34 participants), Acetazolamide 125mg (33 participants), and budesonide 200 mcg (33 participants).

The intervention code will be prepared by Advantage Pharmaceutical using a computer-generated random sequence, and then placed in sealed opaque envelopes unavailable to the study administrators who enroll the patients. Allocation of randomized, blinded study capsules will occur on site at the baseline altitude on a first-come, first-served basis before each participant is identified in order to minimize bias. Success of blinding will be evaluated with a best guess of the intervention question, as well as a statistical evaluation of baseline characteristics to assess for an imbalance in the random allocation of study capsules. A sealed unblinding envelope with the randomization codes will be held by a researcher at BAR as well as a non-study affiliated physician at Stanford University Hospital in the event of an allergic reaction or need for medical intervention.

A word about meals and accommodations: Both Owens Valley Lab and Barcroft Station have a full time chef on staff all year-long who prepare meals for those staying at their respective stations. There are a wide range of options, as it is a full kitchen, with vegetarian, vegan, and normal diet options. Meals are served buffet- style with participants able to eat what they like, and as much as they like. Although meals vary on a daily basis, an average dinner meal might be approximately 2,500 calories and include pasta, meatballs, salad, garlic bread, soup, and steamed vegetable options. If the options for the day are not suiting, the chef can discuss individually with the participant other options. Standard breakfasts include cereals, eggs, sausage, toast, oatmeal, etc. Standard lunches are usually sack-lunch varieties and are often sandwich options with fruit and other snacks. Throughout the day the "snack" portion of the kitchen is open with fruit, sandwich supplies, assortment of bars, chips, etc. Participants are encouraged to bring their own snacks if they have their own snack preferences for hiking. The stations ask that participants assist in cleaning up after themselves as much as possible. No drugs or alcohol are allowed. Accommodations: All participants will be provided with accommodations at both sites and will only be required to bring their own bedding (ie. sleeping bag) and towels. A single twin bed will be provided, arranged alone or as a bunk with no greater than 8 people per co-ed room. If participants would rather camp outside, that is also permitted.

Showers and toilets are available.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female
2. Sea level-dwelling hikers
3. Between ages 18-65

Exclusion Criteria:

1. History of allergy to acetazolamide or budesonide (or other corticosteroids)
2. Taken NSAIDs, acetazolamide, or corticosteroids in the one week prior to study enrollment.
3. Hazardous medical conditions which precludes the ability to moderately hike to high altitude including: sickle cell anemia, asthma, or COPD, severe anemia, or severe coronary arterial disease.
4. Pregnancy or suspected pregnancy.
5. Participants who are younger than 18 years of age and more than 65
6. Sleep above 4'000 elevation in the preceding 1 week.
7. History of asthma or COPD
8. Current symptoms of an acute upper respiratory illness.
9. Unable to complete a moderately strenuous hike at high altitude.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, MD, Principal Investigator — Stanford University
Locations (1):
- Owens Valley Lodge - White Mountain Research Station, Bishop, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lipman GS, Pomeranz D, Burns P, Phillips C, Cheffers M, Evans K, Jurkiewicz C, Juul N, Hackett P. Budesonide Versus Acetazolamide for Prevention of Acute Mountain Sickness. Am J Med. 2018 Feb;131(2):200.e9-200.e16. doi: 10.1016/j.amjmed.2017.05.034. Epub 2017 Jun 28. PMID 28668540

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Budesonide | Acetazolamide | Control
Started | 33 | 35 | 35
Completed | 33 | 35 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Acetazolamide | Control | Total
Number analyzed (Participants) | 33 | 35 | 35 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10) | 33 (9) | 32 (7) | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 21 | 48
  Male | 18 | 23 | 14 | 55
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 35 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Mountain Sickness
Description: Number of participants with acute mountain sickness (AMS) by Lake Lousie Questionnaire (LLQ)
Time Frame: 24 hours
Measure: Number; unit: Count of participants
Arm/Group | Budesonide | Acetazolamide | Control
Number analyzed (Participants) | 33 | 35 | 35
Count of participants | 24 | 22 | 15

2. Secondary Outcome: Number of Participants With Severe Acute Mountain Sickness
Description: Number of participants with severe acute mountain sickness (AMS) by Lake Lousie Questionnaire (LLQ) (score > 5).
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide | Acetazolamide | Control
Number analyzed (Participants) | 33 | 35 | 35
Participants | 18 | 11 | 19

3. Secondary Outcome: Oxygen Saturation
Description: measurement of oxygen saturation (%) by finger tip pulse oximeter.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Budesonide | Acetazolamide | Control
Number analyzed (Participants) | 33 | 35 | 35
percent saturation | 88.6 (4.1) | 88.1 (3.8) | 86.4 (5)

ADVERSE EVENTS:
Arm/Group | Budesonide | Acetazolamide | Control
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes